CLINICAL TRIAL: NCT05397366
Title: Comparison of Task Specific Training Vs Neurodevelopmental Training Along With Conventional Therapy for Upper Limb Motor Function Among Chronic Stroke Patients
Brief Title: Comparison of TSTVs NT Along With Conventional Therapy for Upper Limb Motor Function Among Chronic Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DPT/Batch-Fall17/510
Record Dates: First submitted 2022-05-10; First posted 2022-05-31 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Task Specific Training (Experimental): Using Task Specific Training
  Interventions: Diagnostic Test: Task Specific Training
- Neurodevelopmental Training (Experimental): Using Neurodevelopmental Training
  Interventions: Diagnostic Test: Neurodevelopmental Training

INTERVENTIONS:
Diagnostic Test: Task Specific Training — Group A will be given Task Specific protocol with routine physical therapy treatment for 45 mins on the upper limb for 3 days a week for a period of 12 weeks.
  This Task Specific protocol will include different exercises like, do the polishing of the table top , can perform arm cradling, can supinate and pronate the cylindrical object with arm , while pushing the cylindrical object can extend the wrist , can reach forward to touch or to pick an object , can bend side ways to pick the object and place it on the table in front , can pour the 1/2cup of water to the wide jar that is held by the patient in other hand , patient can comb his hair , patient can drink and eat independently , can lift the jar and bring it close to lips , can pick up pen by using thumb and two fingers , can do the stacking checkers , can throw a ball into the basket , can push the ball on wall from front and side.
  Arms: Task Specific Training
Diagnostic Test: Neurodevelopmental Training — Group B will receive the Neurodevelopmental protocol with the routine physical therapy for 45 mins on the upper limb 3 times a week for period of 12 weeks. The intervention will be performed by the trained physical therapist.
  This Neurodevelopmental protocol will include different exercises like , patient should sit while bearing weight , patient can do self-overhead movements with hand clasped , while holding the gymnastic ball reach forward and overhead position while sitting , weight bearing while plantigrade or quadruped position , while sitting or standing can move the ball in forward , backward and sideways.
  Arms: Neurodevelopmental Training

SUMMARY:
Comparison of Task Specific Training Vs Neurodevelopmental Training Along with Conventional Therapy for Upper Limb Motor Function Among Chronic Stroke Patients

DETAILED DESCRIPTION:
To compare Task Specific Training versus Neurodevelopmental Training along with conventional therapy for upper limb motor function among chronic stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Chronic ischemic stroke patients( after 3 months of stroke ).(41)
* Patients from both gender.(42)
* Patients of around age of 45-65.(43)
* Patient with limb spasticity equal to 2 or less than 2 on modified ash worth scale.(44)
* Patient with good cognitive function minimum 20 or more on Mini Mental State Examination (MMSE).(45)

Exclusion Criteria:

* Patients with history of the recurrent stroke.(41)
* Patient with fracture or dislocation of upper limb.(46)
* Patient with any peripheral vascular disease (47)
* Patient with any comorbid neurological disease like Parkinsonism, epilepsy, multiple sclerosis and spinal cord injury.(21)
* Patient with skin discoloration, skin ulcers and skin allergy.(48)

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2022-05-31 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Neurodevelopmental Training | 6 Months
  37 will receive Neurodevelopmental treatment is based on the premise that the presence of normal postural reflex mechanisms is fundamental to a motor skill's performance. Mini mental state examination test

SECONDARY OUTCOMES:
Task Specific Training | 6 Months
  37 will receive Task specific training is a type of exercise treatment involving repeated practise with your affected arm/hand. Wolf Motor Function Test (WMFT)

CONTACTS AND LOCATIONS:
Locations (1):
- Shadman Medical Centre Chaudhry Muhammad Akram Teaching and Research Hospital University of Lahore Teaching Hospital Services Hospital Lahore General Hospital Bashir Neuro Supine Institute, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No